CLINICAL TRIAL: NCT04012606
Title: A Phase III Randomized, Double-Blind, Placebo-controlled Study of Platinum(Cisplatin or Carboplatin) Plus Etoposide With or Without Toripalimab as First Line Therapy in Patients With ExtensiveStage Small Cell Lung Cancer
Brief Title: Toripalimab in Combination With Platinum Plus Etoposidein Patients With Extensive-Stage Small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JS001-028-III-SCLC
Record Dates: First submitted 2019-07-05; First posted 2019-07-09 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TORIPALIMAB (Experimental)
  Interventions: Drug: TORIPALIMAB INJECTION(JS001 ) Carboplatin Cisplatin Etoposide Placebo
- Chemotherapy (Active Comparator)
  Interventions: Drug: TORIPALIMAB INJECTION(JS001 ) Carboplatin Cisplatin Etoposide Placebo

INTERVENTIONS:
Drug: TORIPALIMAB INJECTION(JS001 ) Carboplatin Cisplatin Etoposide Placebo — TORIPALIMAB INJECTION(JS001 ) or Placebo combined with chemotherapy, 240mg/6ml/vial, Q3W,up to 2 years of treatment.

SUMMARY:
This is a phase III, multicenter, double-blinded, placebo-controlled study of platinum（Cisplatin or Carboplatin） plus etoposide with or without toripalimab as first Line therapy in patients with extensive stage small cell lung cancer.

The purpose of this study is to evaluate the safety and efficacy of toriplimab in combination with platinum（Cisplatin or Carboplatin） plus etoposide in treatment naive extensive stage small cell lung cancer.

Participants will receive asigned study treatment until progressive disease (PD) as assessed by the investigator using Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1).

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years , male or female;
2. Histologically or cytologically confirmed ES-SCLC (per the Veterans Administration Lung Study Group (VALG) staging system
3. ECOG PS 0~1;
4. No prior treatment or immunocheckpoint inhibitors for ES-SCLC;
5. Treatment-free for at least 6 months since last chemo/radiotherapy, among those treated (with curative intent) with prior chemo/radiotherapy for limited-stage SCLC；
6. Patients with asymptomatic brain metastases who have received previous treatment
7. Has provided tumor tissue samples
8. Estimated survival time ≥8 weeks;
9. There is at least one measurable lesion that conforms to RECIST criteria v1.1.For lesions that have received previous radiation therapy, the lesion can only be included in the measurable lesion if the disease progression is clear after radiotherapy and the lesion is not the only measurable lesion.
10. Before the first dose of the study drug, it should have appropriate organ function, and the laboratory test value should meet the protocol.
11. Has adequate hematologic and end organ function

Exclusion Criteria:

1. Prior systemtic treatment for ES-SCLC;
2. Prior treatment with any CD137 agnist or immunocheckpoint inhibitors.
3. Subjects with active or untreated central nervous system (CNS) tumor metastasis;
4. Spinal cord compression not definitively treated with surgery and/or radiation or previously diagnosed and treated spinal cord compression without evidence that disease has been clinically stable for ≥ 1 week prior to randomization
5. Cancerous meningitis;
6. Uncontrolled or symptomatic hypercalcemia;
7. Other malignant tumors within 5 years prior to the first dose of study treatment
8. Subjects with any active, known or suspected autoimmune disease;
9. History of idiopathic pulmonary fibrosis, drug-induced pneumonitis,or evidence of active pneumonitis .
10. Subjects who received major surgery within 28 days prior to enrollment or were not fully recovered from prior surgery;
11. Significant cardiovascular disease, such as New York Heart Assoc

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 442 (Actual)
Dates: Start 2019-07-23 (Actual); Primary Completion 2023-04-20 (Actual); Study Completion 2023-04-20 (Actual)

PRIMARY OUTCOMES:
PFS (Progression Free Survival) by investigator | Approximately 2 years
  Progression free survival (PFS) evaluated by investigators according to the response evaluation criteria in solid tumors (RECIST 1.1)
Overall suvival (OS) | Approximately 2.8 years
  Overall suvival (OS)

SECONDARY OUTCOMES:
PFS (Progression Free Survival) per RECIST1.1 as Assessed by BIRC (Blinded Independent Review Board） | Approximately 2 years
  PFS evaluated by the Blinded Individual Review Committee (BIRC) based on RECIST1.1 criteria;
ORR (Objective Response Rate) | Approximately 2 years
  Objective response rate (ORR) evaluated by investigators and BIRC based on RECIST1.1;
DOR (Duration of Response) | Approximately 2 years
  Duration of response (DOR) evaluated by investigators and BIRC based on RECIST1.1;
DCR (Disease of Response) | Approximately 2 years
  Disease control rate (DCR) evaluated by investigators and BIRC based on RECIST1.1;
TTR (Time to Response) | Approximately 2 years
  Time to response (TTR) evaluated by investigators and BIRC based on RECIST1.1;
OS (Overall Survival) rate | Approximately 2 years
  OS rates at 1 and 2 years
Incidence of AEs/SAEs | Approximately 2 years
  Adverse events (AEs) ; serious adverse events (SAEs); abnormal value of Lab test according to NCI-CTCAE V5.0
PFS (Progression Free Survival) Rate | Approximately 1year
  PFS rates at 6-month（inestigators and BICR） and at 1-year

CONTACTS AND LOCATIONS:
Locations (1):
- Ying Cheng, Changchun, China

REFERENCES:
- [Derived] Cheng Y, Zhang W, Wu L, Zhou C, Wang D, Xia B, Bi M, Fu X, Li C, Lv D, Zhao Y, Chen G, Yi T, Huang J, Li M, Yang R, Huang X, Wang Y, Zhang M, Pan Y, Sun Y, Hu S, Zhang X, Zhou M, Fang J, Jin F, Liu Y, Li Y, Zhang Z, Hu J, Liu L, Wang R, Li Y, Gu K, Ding C, Fan Q, Zhang G, Chen Y, Jiang L, Zheng WE, Chen S, Huang C, Han Z, Yang H, Wang J, Wang B, Wu H, Bao Y, Li M, Luo X, Gu S, Yu W, Xu K, Zhang S, Yu J. Toripalimab Plus Chemotherapy as a First-Line Therapy for Extensive-Stage Small Cell Lung Cancer: The Phase 3 EXTENTORCH Randomized Clinical Trial. JAMA Oncol. 2025 Jan 1;11(1):16-25. doi: 10.1001/jamaoncol.2024.5019. PMID 39541202